CLINICAL TRIAL: NCT04141748
Title: Comparative Effectiveness of Socket Casting Methods: Improving Form and Fit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); INAIL (Istituto Nazionale per L'Assicurazioni contro gli Infortune sul Lavoro) (Unknown); University of Washington (Other)
Responsible Party: Principal Investigator, Steven Gard, Associate Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: W81XWH1910835
Record Dates: First submitted 2019-10-21; First posted 2019-10-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lower Limb Amputation
Keywords: shape capture; prosthetic sockets

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, assessor-blinded, cross-over study
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand Casting (Active Comparator): hand cast will be taken using a circumferential plaster of Paris or fiber glass wrap of the residual limb with the subject in a seated position
  Interventions: Procedure: Hand Casting
- standing hydrostatic pressure casting with a water cylinder (Active Comparator): hand cast will be taken using a circumferential plaster of Paris wrap of the residual limb with the subject in a seated position. The residual limb is then placed into the Symphonie Aqua System while in a weight bearing standing position.
  Interventions: Device: Symphonie Aqua SystemTM

INTERVENTIONS:
Device: Symphonie Aqua SystemTM — a water filled cylinder that can be pressurized around the residual limb to support body weight
  Arms: standing hydrostatic pressure casting with a water cylinder
Procedure: Hand Casting — plaster of Paris or fiberglass bandages are wrapped around the residual limb
  Arms: Hand Casting

SUMMARY:
The overall objective is to compare hand casting to standing hydrostatic pressure casting using a water cylinder in persons with lower limb amputation. Our overall hypothesis is that standing hydrostatic pressure casting with a water cylinder will lead to more consistent and efficient residual limb shape capture and improved initial socket fit and comfort compared to hand casting.

DETAILED DESCRIPTION:
One of the most important components of restoring function in persons with lower limb amputation is the precise fitting of the prosthetic socket to the residual limb. However, this is challenging because the residual limb is dynamic in shape and volume. Additionally, prosthetic socket fabrication processes influence socket fit. These processes typically consist of residual limb shape capture, positive mold rectification, initial diagnostic socket fitting, and definitive prosthesis delivery. The most prevalent residual limb shape capture method involves a negative wrap cast in a non-weight bearing position and manual manipulation of the cast to conform to the residual limb shape. With this technique it is challenging to accurately capture the bony contours and distribute pressure evenly around the residual limb. To improve shape capture, techniques that rely less on manual manipulation by the prosthetist, such as standing hydrostatic pressure casting with a water cylinder have been developed. Given the use of physics to shape the residual limb, it has been proposed that pressure casting results in better fitting and more comfortable sockets, however this has not yet been demonstrated. The overall objective is to compare hand casting to standing hydrostatic pressure casting using a water cylinder in persons with lower limb amputation. Our overall hypothesis is that standing hydrostatic pressure casting with a water cylinder will lead to more consistent and efficient residual limb shape capture and improved initial socket fit and comfort compared to hand casting.

ELIGIBILITY:
Inclusion Criteria:

* unilateral lower limb amputation (transtibial and transfemoral)
* current prosthesis users

Exclusion Criteria:

* poor residual limb sensation
* a superficial neuroma that is painful to pressure
* an open sore on the residual limb
* a residual limb circumference or body weight that exceeds the size or weight limits of the Symphonie Aqua SystemTM (i.e., >58cm and 170kg for persons with transtibial amputation and >78cm and 170kg for persons with transfemoral amputation
* persons who are unable to stand for the 4-6 minutes required for casting (e.g. persons with bilateral amputations).
* persons with new amputations (i.e., have been an amputee for less than 1 year)
* persons with transfemoral amputation who have a known silicone allergy or a femur length less than 5 inches

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Socket Comfort Score | at study completion, 1 month
  Score from 0-10, with 0 being the least comfortable socket and 10 being the most comfortable socket

SECONDARY OUTCOMES:
Cast/Socket volume | at every study visit, up to 1 month
  digitized volume and shape of cast and socket
Procedure time | at every study visit, 1 month
  Time to cast, rectify and fit the socket
Socket Fit | at study completion, 1 month
  checklist will be used to assess fit of socket
Socket preference | at study completion, 1 month
  subject's preference for socket to continue wearing

CONTACTS AND LOCATIONS:
Overall Officials: Steven Gard, PhD, Principal Investigator — Northwestern University
Locations (3):
- United States (2):
  - NUPOC, Chicago, Illinois
  - Minneapolis VA Heath Care System, Minneapolis, Minnesota
- INAIL, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data generated by the funded research will be made available to the research community and to the public under the auspices of the PI. Prior to sharing, data will be de-identified and redacted to reduce the risk of subject identification.
Time Frame: Data will be shared after acceptance for publication of the main findings from the final dataset.
Access Criteria: The PI will share data upon request with anyone via a unique link to a file or folder within Northwestern Box. A data-sharing agreement will be used to ensure that the data is only used for the purpose described, users acknowledge the data source in any use of the data, agree to provide the PI with copies of any presentation or publication that uses the data, prohibit sharing of the data with others without those parties having their own data use agreement, and prohibit manipulation of data for the purposes of identifying subjects.

REFERENCES:
- [Derived] Fatone S, Gravely A, Cutti AG, Hansen AH, Gard SA; Residual Limb Shape Capture Group. Randomized crossover trial of hand and hydrostatic casting for custom lower limb prosthetic sockets: Assessing socket comfort and fabrication time. PLoS One. 2025 Nov 21;20(11):e0337185. doi: 10.1371/journal.pone.0337185. eCollection 2025. PMID 41270063

DOCUMENTS (1):
  • Informed Consent Form (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT04141748/ICF_000.pdf